CLINICAL TRIAL: NCT06587230
Title: Building Teachers Mental Health Skills to Support Students With Mental Health Needs in Elementary and Middle Schools in North Carolina: Program Implementation and Prospective Data Collection
Brief Title: Teachers Leading the Front Lines - North Carolina (Tealeaf-NC)
Acronym: Tealeaf-NC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Darjeeling Ladenla Road Prerna (Unknown); Broadleaf Health and Education Alliance (Other); University of Colorado, Denver (Other); Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 24-1034
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Child Behavior; Mental Health Issue; Psychosocial Functioning; Depression; Anxiety
MeSH Terms: conditions — Child Behavior; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a two-arm, clustered trial evaluating the program implementation of the intervention (Tealeaf) that will be compared to an active comparator (RE-SEED). Schools will be randomized into either the full intervention or a lower-resourced version of the intervention. It is noted that schools are more willing to participate in an intervention trial if they will receive some benefit from their participation, leading to having a lower-resourced comparator rather than a true control comparator. Additionally, the active comparator ethically allows for identified children in need of care to have more resources than if no intervention occurred. Schools, teachers, and students will be followed prospectively with data collection at regular intervals.
Who Masked: Outcomes Assessor
Masking Description: Participants will not be blinded; children must assent, and parents consent, to receive mental health care and teachers will be aware they are delivering care. One research assistant (RA) and staff mental health clinician will not be blinded to observe teachers' fidelity. Otherwise, personnel are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tealeaf (Experimental): Teachers in the Tealeaf arm receive in-depth training and regular supervision and coaching from the study team.
  Interventions: Behavioral: Teachers Leading the Frontlines
- RE-SEED (Active Comparator): Teachers in the RE-SEED arm receive much less in-depth training. The study team does not provide supervision allowing only the school counselor to provide supervision.
  Interventions: Behavioral: Responding to Students' Emotions Through Education

INTERVENTIONS:
Behavioral: Teachers Leading the Frontlines — 1. During 3-day training, Knowledge and attitudes toward child mental health care are measured pre-training, post-training, and post-intervention.
  2. The teachers select students whom they believe have the highest mental health needs to receive care.
  3. Teachers analyze chosen students' symptoms.
  4. Teachers analyze students' behavior with the AABC Chart.
  5. Teachers develop a targeted response using a behavior plan called the 4Cs plan (Cause, Change, Connect, and Cultivate). In the 4Cs, teachers select therapeutic techniques to deliver from a menu of evidence-based therapeutic options for each category of behavior.
  6. Throughout the year, teachers receive supervision through monthly site visits supplemented by as-needed telephone and digital discussions to guide their care from the study team. Teachers encourage the use of the 4Cs plan at home.
  Other Names: Tealeaf
  Arms: Tealeaf
Behavioral: Responding to Students' Emotions Through Education — All processes for RE-SEED are the same as in Tealeaf except...
  1. Teachers receive only 1 day of training
  2. The study team does not provide supervision to the teachers, allowing only the school counselor to provide supervision
  This less resource-intensive approach will allow for an ethical comparator to Tealeaf, where the schools would like for teachers to have some skills to support identified students.
  Other Names: RE-SEED
  Arms: RE-SEED

SUMMARY:
Purpose: The purpose of this research is to pilot test a novel, alternative, potentially sustainable system of teacher-delivered, task-shifted child mental health care.

Participants: ~300 estimated

Procedures: This is a RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) guided, mixed methods, clustered evaluation of Tealeaf-NC's Reach, Adoption & Implementation (Primary Outcomes, implementation-based), as well as evaluating for preliminary indicators of Effectiveness & Maintenance (Secondary Outcomes, clinically-based).

DETAILED DESCRIPTION:
Addressing children's mental health is a critically important health challenge. Twenty percent of all children suffer from significant mental health concerns, most of whom will remain unrecognized, unsupported, and affected throughout their lives. Such wide differences between mental health needs and care access are often called the "care gap". More recently, a youth mental health crisis emerged alongside the COVID-19 pandemic. The adverse impact of the pandemic has led to youth mental health prevalence increasing up to 40% in some global regions, which is double the pre-pandemic rate, while available professional mental health human resources have not changed, leading to an even wider care gap. As urgent solutions are needed, alternative systems of care and support may address this urgent need in a more timely fashion than expanding traditional care systems would.

The overarching goal of this study is to address the youth mental health crisis by providing evidence that high-quality, alternative, sustainable child mental health care may improve youth mental health symptoms. This proposal aims to pilot a novel, alternative, potentially sustainable system of teacher-delivered, task-shifted child mental health care. In North Carolina, USA, the investigators will pilot Teachers Leading the Frontlines - Mansik Swastha [Mental Health in Nepali] (Tealeaf). Created in Darjeeling, India, Tealeaf centers on training and supervising elementary school teachers to deliver "education as mental health therapy" (Ed-MH) to children (ages 5-12). Ed-MH is the investigators' novel, task-shifting, therapy modality that minimizes the time teachers need to deliver care by fitting it into their work. In Ed-MH, teachers use evidence-based therapeutic techniques adapted for use in their existing interactions with students in need (e.g., while teaching) and streamlined for care for any diagnosis ("transdiagnostic").

The investigators' rationale stems from two trials in Darjeeling where the mental health symptoms of children in Tealeaf improved from clinical to neurotypical. The investigators specifically aim to determine if teachers can deliver Tealeaf with fidelity, with positive acceptability & feasibility for stakeholders, and leading to preliminary indicators of improved child mental health outcomes. Guided by the RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) public health framework, the investigators hypothesize that a pilot of Tealeaf clustered at the school level will show that:

1. Teachers can deliver Tealeaf (task-shifted mental health care fitted into their work) with higher fidelity than the active comparator, and stakeholders (teachers, students, parents, principals) will find Tealeaf more acceptable & feasible than the active comparator (Reach, Adoption, Implementation; Primary Outcomes).
2. Tealeaf will show early signs of greater impact on children's 1) mental health symptoms, 2) academic achievement, and 3) school attendance versus a comparator (Effectiveness, Maintenance; Secondary Outcomes).

Researchers will compare Tealeaf with an active comparator, RE-SEED (Responding to Students' Emotions through Education), to see if a lower-resourced version of Tealeaf is viable and/or has an impact.

Tealeaf has six components implemented over a school year:

1. Teachers first complete three days of training, delivered by a mental health professional (e.g. psychiatric social worker, psychologist, or psychiatrist).
2. Teachers use a study-specific tool, the Behavior Type and Severity Tool (BTST), to systematically capture their impression of each student in their class. Using their judgment, aided by the BTST, teachers select students whom they believe have the highest mental health needs to receive care.
3. Teachers observe chosen students' symptoms with the Strengths and Difficulties Questionnaire. (If the child has a positive total or subscale score, they are eligible for the study. The target enrollment of ~2 students per teacher based on estimated prevalence and teacher feedback on a feasible case load).
4. Teachers understand students' behavior using the Activating Event, Automatic Thought/or Feeling, Behavior, and Consequence Chart (AABC Chart) and the Themes of the AABC Chart tool. These tools are similar to the Antecedent, Behavior, and Consequences (ABC) Chart from Cognitive Behavior Therapy (CBT).
5. Teachers develop a targeted response using a plan called the 4Cs (Cause, Change, Connect, and Cultivate) plan. The chosen care framework for addressing behavior and mental health and that the 4Cs was modeled on are behavior plans (not manualized care). They align with how teachers already individualize teaching to students' needs. The 4Cs' goal is to improve mental health through and in addition to learning, whereas typical behavior plans solely target improved learning. In the 4Cs, teachers select therapeutic techniques to deliver from a menu of evidence-based therapeutic options for each category of behavior. Ed-MH adapts Cognitive Behavior Play Therapy (CBPT) and Dialectical Behavior Therapy (DBT) measures for classroom delivery. Based on CBT, CBPT is accessible to children <10 years old using both talk and play therapy. There are two chosen areas of therapeutic focus for teachers. 1) Behavioral activation and self-regulation are guided by the teachers as they occur in the classroom. 2) Cognitive restructuring is incorporated through traditional means (AABC Chart).
6. The remainder of the school year is dedicated to the development of therapeutic relationships and the delivery of therapeutic interactions and skills practice. Revisions to the 4Cs plan are made based on each child's progress. As a key component of task-shifting, teachers receive supervision through monthly site visits supplemented by as-needed telephone and digital discussions to guide their care from the study team. This supervision occurs throughout the year. Trained school counselors can also provide monthly supervision or as needed. Teachers encourage the use of the 4Cs plan at home.

For RE-SEED (active comparator), processes are similar to Tealeaf. The differences are that training is 1-day such that they receive markedly less in-depth knowledge, and the study team does not provide supervision, allowing only the counselor to provide supervision. This less resource-intensive approach will allow for an ethical comparator to Tealeaf, where schools would like for teachers to have some skills to support identified students as part of their willingness to participate in research, while also allowing the investigators to begin to understand what impact fewer resources may have versus a full intervention.

Tealeaf and Ed-MH's mechanism of action for improving mental health symptoms is through teachers guiding children to consistently practice coping skills and emotion regulation for long periods (a school day) and in real-time (in moments of concern). Like counselors, Tealeaf teachers help students gain insight and acquire coping skills. Teachers take the therapy activities further, though, by overseeing children practicing coping skills, reinforcing positive behavior, and supporting them in moments of struggle, all in real-time. It is ideally how teachers would work with students as guided by a therapist, but here they determine how to therapeutically respond to a student's mental health needs since therapists are inaccessible. Moreover, as a role model, teachers already play a key role in the social, emotional, and academic development of students and interact with them individually in moments of concern. Ed-MH allows teachers to deliver therapy in shared moments, in real time. Professional and lay counselors, instead, can only reflect from afar on moments the student is willing to share in the office.

A second mechanism of action is through teachers delivering care that can target education symptoms of mental health as seen in India. For example, a student may have poor schoolwork due to anxiety. Their teacher can target their poor schoolwork (the education symptoms of their mental health) and anxiety by improving schoolwork quality (an education intervention) by building their capacity to complete assignments gradually, i.e. exposure therapy (an evidence-based technique). After care, both symptoms improved.

Intervention evidence: Results from 2018 and 2019 pilot Tealeaf trials show that mental health care delivery for children can be shifted to teachers.

1. Teachers (n=19) nominated students (n=36) with moderate accuracy, 72% sensitivity, and 62% specificity, aligned with identification by lay counselors in Low- or Middle- Income Countries (LMIC) and teachers in High-Income Countries (HIC).
2. Teachers (n=19) delivered care with fidelity, on average at or above 60% fidelity to protocol, similar to mental health professionals' fidelity to new therapies.
3. Teachers (n=19) found it feasible to deliver therapy when integrated into their workflow (Ed-MH), citing the choice of therapeutic techniques and the ability to incorporate them into teaching.
4. Teachers, families, and students found it acceptable for teachers to deliver mental health care. Teachers cited flexible care delivery, families cited impact, and students cited being treated well.
5. Children's mental health symptoms improved after receiving Ed-MH from their teachers, an early signal of impact. Symptoms improved on average from clinical to neurotypical, i.e., from the 77th to the 60th percentile baseline to end line on a gold standard measure in 2018 (n=36) and from the 84th to the 68th percentile in 2019 (n=26). While supported children in 2019 had neurotypical symptom levels at the end line, children receiving enhanced usual care (n=188) remained at clinical levels (81st percentile; effect size 0.7) These findings support teachers' delivery of task-shifted, indicated child mental health care that is transdiagnostic and integrated into their work.

Overall, our prior research demonstrates that teacher-delivered transdiagnostic mental health care (Tealeaf inclusive of Ed-MH) may be a potentially efficient, sustainable, and impactful approach. A Type 1 hybrid effectiveness-implementation Tealeaf trial is ongoing in Darjeeling, India.

The investigators' rationale for pilot testing Tealeaf-NC is based on Tealeaf's promising results as there is an urgent need to identify and deliver evidence-based children's mental health interventions to tackle the children's mental health care gap that worsened into a crisis during the COVID pandemic. Of note, Tealeaf skipped over efficacy (lab-like setting) to effectiveness testing (real world), as literature supports skipping efficacy testing of task-shifted mental health care. Task-shifting improves mental health outcomes in lab-like settings and is now recommended to be tested in specific forms (e.g., teacher-delivery) for specific contexts to study its effects in real-world practice. As research evidence takes an average of 17 years to reach clinical practice, and given Tealeaf's promise, the urgent need justifies pilot testing Tealeaf's potential implementation and clinical outcomes in new settings.

ELIGIBILITY:
Inclusion Criteria:

Schools:

* Have been trained in either Tealeaf or RE-SEED in Summer 2024 or 2025 after being randomized programmatically
* Be a school in the State of North Carolina
* Have an eligible principal

Principals:

* >18 years old
* Employed at an enrolled school
* Not suspected or convicted of child-related misconduct or maltreatment

Teachers:

* >18 years old
* Employed at an enrolled school
* Primary teaching responsibility for a single academic class (for a minimum of 1 hour per day and a minimum of 4 days per week) in any grade level Kindergarten to Grade 8
* Not suspected or convicted of child-related misconduct or maltreatment

Counselors:

* >18 years old
* Employed at an enrolled school
* Hold a school counselor position at an enrolled school for at least 10 hours per week
* Not suspected or convicted of child-related misconduct or maltreatment

Students:

* Enrolled in Kindergarten-Grade 8
* Student of an enrolled teacher
* Has a parent or guardian who can provide consent
* Positive/Clinical-level score on the Strengths and Difficulties Questionnaire (SDQ)

Guardians:

* >18 years old
* Guardian of enrolled student

Exclusion Criteria:

* Exclusion criteria will be set as each participant does not meet the inclusion criteria as set for their group.

Ages: 5 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Mean Acceptability of Intervention Measure (AIM) Scores | Month 0, Month 9
  The Acceptability of Intervention Measure (AIM) measures the stakeholder's beliefs about the acceptability of the assigned intervention. Each element is scored from 1 (Completely disagree) to 5 (Completely agree). Mean scores are calculated, with a higher score indicating that the teacher believes the intervention is more acceptable, and a score greater than or equal to 4 indicating positive acceptability.
Mean Intervention Appropriateness Measure (IAM) Scores | Month 0, Month 9
  The Intervention Appropriateness Measure (IAM) measures the stakeholder's beliefs about the appropriateness of the assigned intervention. Each element is scored from 1 (Completely disagree) to 5 (Completely Agree). Mean scores are calculated, with a higher score indicating that the teacher believes the intervention is more appropriate, and a score greater than or equal to 4 indicating the intervention is more appropriate.
Mean Feasibility of Intervention Measure (FIM) Scores | Month 0, Month 9
  The Feasibility of Intervention Measure (FIM) measured the stakeholder's beliefs about the feasibility of the assigned intervention. Each element is scored from 1 (Completely disagree) to 5 (Completely agree). Mean scores are calculated, with a higher score indicating that the teacher believes the intervention is more feasible, and a score greater than or equal to 4 indicating positive feasibility.
Mean Cause Analysis Chart (AABC) Evaluation Checklist Scores | Month 9
  The Cause Analysis Chart (AABC) Evaluation Checklist is a study-specific tool that assists evaluators in scoring the fidelity with which teachers accurately complete the AABC Chart. Mean scores are calculated and can range from 1 (Needs improvement) to 5 (Advanced) with a higher mean score indicating higher fidelity, and an overall mean score greater than or equal to 4 indicating sufficient fidelity.
Mean 4Cs Behavior Plan Evaluation Checklist Scores | Month 9
  The 4Cs Behavior Plan Evaluation Checklist is a study-specific tool that assists evaluators in scoring the fidelity with which teachers accurately complete the 4Cs Behavior Plan. Mean scores are calculated and can range from 1 (Needs improvement) to 5 (Advanced) with a higher mean score indicating higher fidelity, and an overall mean score greater than or equal to 4 indicating sufficient fidelity.
Mean One-on-One Student Interaction Evaluation Tool Scores | Month 9
  The One-on-One Student Interaction Evaluation Tool is a study-specific tool that measures the fidelity with which teachers conduct one-on-one sessions with the student(s). Teachers are rated on six domains on a scale that ranges from 1 (Needs Improvement) to 5 (Advanced). Scores are averaged and rounded to a half point across domains to yield mean scores from 1 to 5 with a mean higher score indicating higher fidelity, and a mean score greater than or equal to 4 indicating sufficient fidelity.
Mean One-on-One Family Interaction Evaluation Tool Scores | Month 9
  The One-on-One Family Interaction Evaluation Tool is a study-specific tool that measures the fidelity with which teachers conduct family interactions. Teachers are rated on six domains on a scale that ranges from 1 (Needs improvement) to 5 (Advanced). Scores are averaged and rounded to a half point across domains to yield mean scores from 1 to 5 with a mean higher score indicating higher fidelity, and a mean score greater than or equal to 4 indicating sufficient fidelity.

SECONDARY OUTCOMES:
Change in Strengths and Difficulties Questionnaire Total Difficulties Score | Month 0, Month 9
  The Strengths and Difficulties Questionnaire is a brief behavioral screening that will measure the mental health of students, and the change in scores will measure the effectiveness of the assigned intervention. The total difficulties score is the summation of 4 subscales: emotional symptoms, conduct problems, hyperactivity/inattention, and peer relationship problems. Each subscale has 5 items scored as "Not True," "Somewhat True," and "Certainly True" yielding a value of 0,1, or 2. (Some items are scored in reverse). The total difficulties score is generated by summing scores from each scale to yield an overall score. The overall score range is from 0-40, with a higher score indicating more difficulties/worse mental health. A bigger decrease in the total difficulties scores will indicate that the intervention is more effective.
Mean Proportion of Attendance | Up to 18 months
  Using the teachers' and school records, the number of days present will be converted to a proportion of days in attendance (due to the varied length of academic school years). These proportions will be compared between arms, and a higher proportion of attendance will indicate a more effective intervention.
Change in Academic Achievement | Up to 18 months
  Using the teachers' and school records, a change in student academic achievement score will be coded from available grades, assessment, discipline and IEP/504 information. A significant change in the positive direction will indicate an effective intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Christina R Cruz, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with The University of North Carolina (UNC).
Time Frame: Data will be available beginning 12 and continuing for 36 months after publication to allow researchers to analyze data and submit for peer review.
Access Criteria: Data will be deposited in UNC Odum Institute's UNC Dataverse, an open-source data repository service for the University of North Carolina at Chapel Hill (UNC) research community and its partners.
URL: https://dataverse.unc.edu/

REFERENCES:
- [Background] van Ginneken N, Tharyan P, Lewin S, Rao GN, Meera SM, Pian J, Chandrashekar S, Patel V. Non-specialist health worker interventions for the care of mental, neurological and substance-abuse disorders in low- and middle-income countries. Cochrane Database Syst Rev. 2013 Nov 19;(11):CD009149. doi: 10.1002/14651858.CD009149.pub2. PMID 24249541
- [Background] van Ginneken N, Chin WY, Lim YC, Ussif A, Singh R, Shahmalak U, Purgato M, Rojas-Garcia A, Uphoff E, McMullen S, Foss HS, Thapa Pachya A, Rashidian L, Borghesani A, Henschke N, Chong LY, Lewin S. Primary-level worker interventions for the care of people living with mental disorders and distress in low- and middle-income countries. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD009149. doi: 10.1002/14651858.CD009149.pub3. PMID 34352116
- [Background] Patel V, Kieling C, Maulik PK, Divan G. Improving access to care for children with mental disorders: a global perspective. Arch Dis Child. 2013 May;98(5):323-7. doi: 10.1136/archdischild-2012-302079. Epub 2013 Mar 9. PMID 23476001
- [Background] Shinde S, Weiss HA, Varghese B, Khandeparkar P, Pereira B, Sharma A, Gupta R, Ross DA, Patton G, Patel V. Promoting school climate and health outcomes with the SEHER multi-component secondary school intervention in Bihar, India: a cluster-randomised controlled trial. Lancet. 2018 Dec 8;392(10163):2465-2477. doi: 10.1016/S0140-6736(18)31615-5. Epub 2018 Nov 22. PMID 30473365
- [Background] Burns BJ, Costello EJ, Angold A, Tweed D, Stangl D, Farmer EM, Erkanli A. Children's mental health service use across service sectors. Health Aff (Millwood). 1995 Fall;14(3):147-59. doi: 10.1377/hlthaff.14.3.147. PMID 7498888
- [Background] Kola L, Kohrt BA, Hanlon C, Naslund JA, Sikander S, Balaji M, Benjet C, Cheung EYL, Eaton J, Gonsalves P, Hailemariam M, Luitel NP, Machado DB, Misganaw E, Omigbodun O, Roberts T, Salisbury TT, Shidhaye R, Sunkel C, Ugo V, van Rensburg AJ, Gureje O, Pathare S, Saxena S, Thornicroft G, Patel V. COVID-19 mental health impact and responses in low-income and middle-income countries: reimagining global mental health. Lancet Psychiatry. 2021 Jun;8(6):535-550. doi: 10.1016/S2215-0366(21)00025-0. Epub 2021 Feb 24. PMID 33639109
- [Background] Liang L, Ren H, Cao R, Hu Y, Qin Z, Li C, Mei S. The Effect of COVID-19 on Youth Mental Health. Psychiatr Q. 2020 Sep;91(3):841-852. doi: 10.1007/s11126-020-09744-3. PMID 32319041
- [Background] Frontiers Production Office. Erratum: The Potential Emergence of "Education as Mental Health Therapy" as a Feasible Form of Teacher-Delivered Child Mental Health Care in a Low and Middle Income Country: A Mixed Methods Pragmatic Pilot Study. Front Psychiatry. 2022 Jan 18;12:838044. doi: 10.3389/fpsyt.2021.838044. eCollection 2021. PMID 35115975
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Wong G, Greenhalgh T, Westhorp G, Buckingham J, Pawson R. RAMESES publication standards: realist syntheses. J Adv Nurs. 2013 May;69(5):1005-22. doi: 10.1111/jan.12095. Epub 2013 Jan 29. PMID 23356726
- [Background] Pawson R, Greenhalgh T, Harvey G, Walshe K. Realist review--a new method of systematic review designed for complex policy interventions. J Health Serv Res Policy. 2005 Jul;10 Suppl 1:21-34. doi: 10.1258/1355819054308530. PMID 16053581
- [Background] Cruz CM, Dukpa C, Vanderburg JL, Rauniyar AK, Giri P, Bhattarai S, Thapa A, Hampanda K, Gaynes BN, Lamb MM, Matergia M. Teacher, caregiver, and student acceptability of teachers delivering task-shifted mental health care to students in Darjeeling, India: a mixed methods pilot study. Discov Ment Health. 2022;2(1):21. doi: 10.1007/s44192-022-00024-z. Epub 2022 Oct 31. PMID 36341156
- [Background] Pearson N, Naylor PJ, Ashe MC, Fernandez M, Yoong SL, Wolfenden L. Guidance for conducting feasibility and pilot studies for implementation trials. Pilot Feasibility Stud. 2020 Oct 31;6(1):167. doi: 10.1186/s40814-020-00634-w. PMID 33292770
- [Background] Arain M, Campbell MJ, Cooper CL, Lancaster GA. What is a pilot or feasibility study? A review of current practice and editorial policy. BMC Med Res Methodol. 2010 Jul 16;10:67. doi: 10.1186/1471-2288-10-67. PMID 20637084
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. Correction to: A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2023 Mar 11;23(1):59. doi: 10.1186/s12874-023-01880-1. No abstract available. PMID 36927764